CLINICAL TRIAL: NCT01652378
Title: Pharmacologic MRI in Cocaine-addiction
Brief Title: Pharmacologic MRI in Cocaine Addiction
Acronym: phMRI
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: STU 122011-052
Record Dates: First submitted 2012-06-12; First posted 2012-07-30 (Estimated); Last update posted 2019-09-09 (Actual); Status verified 2019-09

CONDITIONS: Cocaine Dependence
Keywords: cocaine addiction; neuroimaging; functional magnetic resonance imaging (fMRI)
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Ondansetron; Lidocaine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cocaine-Addicted Participants: Group of participants diagnosed with cocaine dependence
  Interventions: Drug: ondansetron, lidocaine
- Control Participants: healthy control volunteers
  Interventions: Drug: ondansetron, lidocaine

INTERVENTIONS:
Drug: ondansetron, lidocaine — Ondansetron: Ondansetron (0.15 mg/kg) will be administered through the IV line over 15 min at a constant rate of infusion.
  Lidocaine: Lidocaine will be administered as a 2mg/kg initial bolus over 5 minutes followed by a continuous intravenous infusion of lidocaine at a rate of 2mg/kg/hour for 55 min (60 min total infusion).
  Other Names: Zofran, Xylocaine

SUMMARY:
In the proposed study, the investigators will assess the brain response to medication probes the investigators have previously studied with SPECT. The brain response to ondansetron and lidocaine infusions will be measured Arterial Spin Labeling and functional connectivity MRI (fcMRI).

DETAILED DESCRIPTION:
An extensive effort has been mounted to understand the neurobiologic mechanisms involved in the development and persistence of cocaine addiction and tendency to relapse. Although the last two decades have resulted in an explosion in our understanding of the biological mechanisms of reward, establishing the relevance of this knowledge to the addictive process has been problematic. Most importantly, this information has been of limited utility in offering new pharmacologic treatment approaches to addicted patients - particularly those with cocaine addiction. Over the past 15 years our laboratory has published multiple studies using pharmacologic probes to explore the biologic underpinnings of cocaine addiction using single photon emissions computerized tomography (SPECT) technology. More recently, however, functional magnetic resonance imaging (fMRI) has offered several advantages over SPECT and is now a favored approach, e.g. fMRI allows the continuous measurement of neural responses rather than a very limited time period with SPECT (1-3 minutes every 48 hours). Using fMRI [including both ASL (Arterial Spin Labeling) and fcMRI (functional connectivity], the neural response can be measured throughout the 60 min that follows infusion, allowing identification and capture of the maximal brain response period that may occur at any time during this 60 min. In the proposed study, we will assess the brain response to two of the probes (scopolamine and lidocaine) we have previously studied with SPECT.

ELIGIBILITY:
Inclusion Criteria:

* Cocaine dependence (cocaine patients)
* identify cocaine as their present primary drug of use
* Patients must have used cocaine within the previous 4 weeks (by patient history) and be abstinent for at least 1 week.
* No drug dependence (healthy control population).

Exclusion Criteria:

* Other medical or psychiatric disorders that may effect neural functioning.
* Medications that may effect brain functioning

Ages: 21 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Subjects with cocaine addiction will be recruited from patients requesting treatment for addiction at the Dallas VA Medical Center and Homeward Bound,Inc. Recently using cocaine patients and healthy controls will be recruited from flyers and internet ads.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2012-08; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
blood-oxygen-level-dependent contrast (BOLD) | 60 minutes after drug infusion
  change in BOLD response to drug infusion (ondansetron, lidocaine).

CONTACTS AND LOCATIONS:
Overall Officials: Bryon Adinoff, M.D., Principal Investigator — UT Southwestern Medical Center at Dallas
Locations (1):
- UT Southwestern Medical Center at Dallas, Divison on Addictions, Dallas, Texas, United States